CLINICAL TRIAL: NCT03746886
Title: Lipids and Other Bioactive Compounds of Human Breast Milk and Infant Formulas.
Brief Title: Lipids and Other Bioactive Compounds of Human Breast Milk
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, Kaisa Linderborg, Associate Professor, University of Turku
Other Study IDs: Korvike
Record Dates: First submitted 2018-11-07; First posted 2018-11-20 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Breast Milk Collection
Keywords: breast milk; lipids; bioactive compounds; infant formula
MeSH Terms: conditions — Breast Milk Expression | interventions — Milk

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Human breast-milk samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast-feeding women: A single breast-milk sample will be collected from 20 women who breast-feed their child (0-6 months old).
  Interventions: Other: Breast-milk

INTERVENTIONS:
Other: Breast-milk — A single breast-milk sample will be collected from 20 women. Milk samples will be pooled for analysis.

SUMMARY:
The biochemical differences in the composition of breast milk and formula have not been profoundly established in all compound groups. Increased understanding of breast milk composition, the normal variation of various bioactive compounds and their levels is required to be able to develop formulas better corresponding the breast milk, and ensure the optimal development of also the formula-fed babies.

ELIGIBILITY:
Inclusion Criteria:

* breast-fed child was born full-time and is healthy.
* age of the breast-fed child is 0-6 months

Exclusion Criteria:

* breast-fed child was born prematurely (gestation week <37)

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Self-representation
Study Population: 18-45 years old women who breast-feed their 0-6 months old child
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Relative proportions (%) of regioisomers within selected molecular species (acyl carbon number:number of double bonds 50:1 and 52:2) in triacylglycerols. | 11/2018-12/2019
  Isolation of lipids from the milk with solvent extraction. Isolation of triacylglycerols with solid phase extraction. Negative ionization of the triacylglycerols with ammonia. Selection of the molecular weight species in the first quadruple of the MS/MS. Fragmentation of the selected ions with argon. Separation of the fragment ions in the second quadrupole of the MS/MS. Calculation of the relative proportions of regioisomers with a computer software.
Relative proportions (%) of fatty acids in triacylglycerols of human milk. | 11/2018-12/2019
  Isolation of lipids from the milk with solvent extraction. Isolation of triacylglycerols with solid phase extraction. Quantitation with gas chromatograph coupled with flame ionization detector in relation to external standards.
Quantity (mg/ml) of lipid soluble compounds in triacylglycerols of human milk. | 11/2018-12/2019
  Isolation of lipids from the milk with solvent extraction. Gravimetric analysis of the lipids.

CONTACTS AND LOCATIONS:
Overall Officials: Kaisa M Linderborg, PhD, Principal Investigator — University of Turku
Locations (1):
- Department of Biochemistry, University of Turku, Turku, Finland

IPD SHARING:
Plan to Share IPD: Undecided